CLINICAL TRIAL: NCT06250699
Title: A Single Center Randomized Controlled Study on the Promotion of Rapid Recovery Through Tubeless Laparoscopic Adrenalectomy
Brief Title: A Single Center Randomized Controlled Study on the Promotion of Rapid Recovery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhe Meng (Other)
Responsible Party: Sponsor-Investigator, Zhe Meng, Deputy chief physician, Zhongnan Hospital
Organization: Zhongnan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023231
Record Dates: First submitted 2024-01-28; First posted 2024-02-09 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Nonfunctional Adrenal Cortex Adenoma; Primary Aldosteronism; Cushing Syndrome
Keywords: tubeless; laparoscopic adrenalectomy; rapid recovery
MeSH Terms: conditions — Hyperaldosteronism; Cushing Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- no tube (Experimental): no drainage tube after laparoscopic adrenalectomy
  Interventions: Procedure: Tubeless laparoscopic adrenalectomy
- Drainage tube (Experimental): tube drainage after laparoscopic adrenalectomy
  Interventions: Procedure: Drainage tube

INTERVENTIONS:
Procedure: Tubeless laparoscopic adrenalectomy — No drainage tube placed after laparoscopic adrenalectomy
  Arms: no tube
Procedure: Drainage tube — Placing drainage tubes after laparoscopic adrenalectomy
  Arms: Drainage tube

SUMMARY:
The goal of this clinical trial is to exploring the role of tubeless after adrenalectomy surgery. The main questions it aims to answer are:

1. The safety of tubeless laparoscopic adrenalectomy；
2. The role of tubeless therapy in rapid recovery after adrenalectomy surgery Participants will be randomly divided into two groups: the non drainage group and the drainage group after laparoscopic adrenal surgery, and their pain, first time out of bed, and intestinal recovery time will be observed.

DETAILED DESCRIPTION:
The design type of this study is a prospective single center randomized controlled study, with a plan to recruit 200 patients who underwent laparoscopic adrenalectomy for the study. The intervention measures mainly include whether to indwelling drainage tubes. Prior to the start of the trial, our center had performed laparoscopic adrenalectomy on 89 patients without any obvious retroperitoneal fluid accumulation, redness, swelling, or fever, and the recovery was smooth. Step 1 of the research: Select patients who meet the criteria for laparoscopic adrenalectomy Step 2: Sign informed consent form Step 3: Randomly draw lots and divide them into two groups: no tube group (experimental group of 100 cases) and indwelling drainage tube group (control group of 100 cases) Step 4: Perform surgical plan according to grouping results Step 5: Test blood routine and ERAS related indicators 1-3 days after surgery Step 6: Follow up adrenal ultrasound at 1 month and 6 months after surgery Step 7: Follow up and analyze data Random plan Use block randomization method, using software SAS9.4 TS1M7, random seed number 2023092311 Observation items and testing time points 1. Test hemoglobin and drainage volume on 1-3 days after surgery Pain score, first time out of bed, intestinal ventilation time, adrenal ultrasound, postoperative fever, wound infection, and other indicators; During the follow-up one month after surgery, the adrenal region color ultrasound should also be tested; 3. During the follow-up examination at 6 months after surgery, ultrasound of the adrenal region should also be detected; Efficacy evaluation criteria and effectiveness evaluation methods: Whether the indwelling drainage tube has a promoting effect on the patient's rapid recovery (such as pain score, first time out of bed, intestinal ventilation time, etc.). Safety evaluation methods mainly include the subject's blood routine and vital signs.

ELIGIBILITY:
Inclusion Criteria:

1. According to the 2022 edition of the Chinese Guidelines for Diagnosis and Treatment of Urological Diseases, patients who meet the surgical indications
2. The patient has signed an informed consent form before joining the clinical trial, and the age at the time of signing the informed consent form is 18-70 years old.

Exclusion Criteria:

1. Patients with complications that seriously affect treatment or quality of life
2. The patient has any physical condition that the researcher believes will affect the clinical status
3. Patients who have placed vascular stents such as heart and cerebrovascular stents within the past year
4. Pregnant or lactating patients

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-01-03 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Pain score | 1-3 days after surgery
  Pain rating scale after laparoscopic adrenalectomy by VAS（visual analog scale for pain ） scale. The score ranges from 1 to 10, and the degree of pain gradually increases.
First time up and about | 1-3 days after surgery
  First time up and about after laparoscopic adrenalectomy
Recovery time of intestinal function | 1-3 days after surgery
  Recovery time of intestinal function after laparoscopic adrenalectomy
Hematoma | 1-3 days after surgery
  Detection of obvious hematoma (Hematoma area> 4cm x 4cm) in the surgical area through color ultrasound. The results are expressed as yes or no.

SECONDARY OUTCOMES:
fever | 1-3 days after surgery
  Does the patient experience fever (The thermometer shows a temperature greater than 37.3 ° C) after laparoscopic adrenalectomy.

CONTACTS AND LOCATIONS:
Overall Officials: meng zhe, Principal Investigator — Wuhan University
Locations (1):
- Zhongnan hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chai S, Pan Q, Liang C, Zhang H, Xiao X, Li B. Should surgical drainage after lateral transperitoneal laparoscopic adrenalectomy be routine?-A retrospective comparative study. Gland Surg. 2021 Jun;10(6):1910-1919. doi: 10.21037/gs-20-829. PMID 34268075
- [Background] Lelli G, Micalizzi A, Iossa A, Fassari A, Concistre A, Circosta F, Petramala L, De Angelis F, Letizia C, Cavallaro G. Application of enhanced recovery after surgery (ERAS) protocols in adrenal surgery: A retrospective, preliminary analysis. J Minim Access Surg. 2024 Apr 1;20(2):163-168. doi: 10.4103/jmas.jmas_319_22. Epub 2023 May 10. PMID 37282440